CLINICAL TRIAL: NCT02066935
Title: Non-adherence to Immunosuppressives in Kidney Transplantation in Brazil: Diagnosis and Associations - ADHERE BRAZIL Multicenter Study
Brief Title: Non-adherence to Immunosuppressives in Kidney Transplantation in Brazil Multicenter Study
Acronym: ADHEREBRAZIL
Status: Completed | Type: Observational
Sponsor: Fundação Instituto Mineiro de Estudo Pesquisa Em Nefrologi (Other)
Collaborators: Hospital das Clínicas de São Paulo - SP (Unknown); Instituto de Urologia e Nefrologia - São José Rio Preto/SP (Unknown); Hospital do Rim/UNIFESP - SP (Unknown); Hospital Israelita Albert Einstein (Other); Hospital de Clinicas da Unicamp - SP (Unknown); Hospital São Francisco de Assis na Providência de Deus - RJ (Unknown); Hospital Universitário UFJF - MG (Unknown); Santa Casa de Juiz de Fora - MG (Unknown); Fundação Prorim Hospital Municipal de São José Joinvile - SC (Unknown); Santa Casa de Porto Alegre - RS (Unknown); Hospital das Clínicas de Porto Alegre - RS (Unknown); Hospital e Maternidade Angelina Caron - SC (Unknown); Hospital Universitário do Maranhão - MA (Unknown); Hospital Walter Cantidio - CE (Unknown); Hospital Ofir Loyola - PA (Unknown); Santa Casa de Misericórdia de Belo Horizonte - MG (Unknown); Hospital São João de Deus - Divinolopis-MG (Unknown); Hospital Antonio Targino- PB (Unknown); University of Brasilia (Other); Hospital Onofre Lopes - RN (Unknown)
Responsible Party: Principal Investigator, Helady Pinheiro, MD, PhD, MD; PhD, Fundação Instituto Mineiro de Estudo Pesquisa Em Nefrologi
Other Study IDs: ADHEREBZ-001
Record Dates: First submitted 2013-10-10; First posted 2014-02-20 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Medication Adherence
Keywords: immunosuppression; medication nonadherence; kidney transplantation
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- kidney transplant patient: Kidney transplanted patients for at least one year
  Interventions: Other: kidney transplant patient

INTERVENTIONS:
Other: kidney transplant patient — kidney transplanted patients for at least one year

SUMMARY:
The purpose of the study are: 1. To estimate the prevalence of non-adherence to immunosuppressants, and to other treatment-related aspects (smoking cessation, alcohol consumption, physical activity, and appointment keeping), in KT recipients among different KT centres across different regions of Brazil; 2. To explore multilevel factors associated to immunosuppressive adherence at the level of patient (socio-demographic, clinical), healthcare provider (patient satisfaction with the interpersonal dimension of care, trust in the transplant team, social support), healthcare organization (composition of the team, operational access, CIM transplant program practice patterns), and healthcare system and policies (perceived financial burden of the treatment regimen, insurance status, barriers to access to the immunosuppressive drugs, Brazilian region);

DETAILED DESCRIPTION:
Kidney transplant (KTx) is considered the best therapeutic option for patients with chronic kidney disease (CKD), based not only on medical reasons, but also on socioeconomic ones1. One of most important determinants of kidney transplants survival is the adherence to immunosuppressive drugs. Adherence may be defined as a patient's behavior agreement regarding the prescribed treatment, including the extent to which a person takes medications, follows a diet and/or implements lifestyle changes as prescribed by health care providers. In the setting of transplantation, a recent consensus conference stated nonadherence (NAd) as "deviation from the prescribed medication regimen sufficient to adversely influence the regimen's intended effect". Risk factors for NAd, have been categorized by the WHO into five dimensions: socioeconomic factors, disease, treatment factors, patient condition and health care team and health system characteristics. 2 Looking at all vascularized transplant recipients, KTx patients are reported like the most non-adherent.3 In Brazil, which is currently the second country in the absolute number of TxR, there are only two studies about prevalence of NAd, lacking in representativeness of the Brazilian scenario4,5. In 2012, 5.385 TxR were performed, but have clear regional differences in that activity: localized mostly in the South and Southeast regions, and performed by big services with high transplant activity transplantation. In this context, the approach of NAd can be fundamental importance in view of their influence on the results.6 The scientific literature recommends to use more than one a method for assessing adherence of the therapeutic regimen. Each method has advantages and disadvantages, and no method is actually considered the gold standard. On the other hand, a combination of measures maximizes accuracy to diagnostic of NAd.7,8 We intent to identify the prevalence of NAd to immunosuppressives in Brazilian kidney transplant patients, by using the more appropriated methodology of triangulation. As secondary objectives we will design the differences between centers and regions of the country as well the risk factors to NAd.

SAMPLE, SETTING AND DATA COLLECTION

Sample, Setting: The sample size was defined based on data from the 2012 Brazilian Registry of Transplant (2012 RBT)6 available by the Brazilian Association of Transplantation (ABTO). The total number of patients transplanted in Brazil from 2000 to 2012 was 59,001 , and 20,504 patients have been registered to be monitored in transplant centers who contribute to that register. Using the OpenEpi stats program, the sample was calculated for studies of population frequency, considering the hypothetical 50% confidence interval of 5% and design effect ranging from 2.0 to 3.0. The obtained sample size ranged from 755 to 1130 patients.

Selection of the centers participating in the study: According to 2012 RTB, there are 123 active transplant center in Brazil, distributed by 22 states, which performed 5.385 KTxs in that year. We will arbitrarily divide the centers in two regions, according to their transplantation activity: Region 1 or high activity, including centers from South and Southeast region, and Region 2 or low / moderate activity accomplishing centers from North, Northeast and Midwest. To ensure representativeness of the characteristics of the centers we will also take in account other characteristics: transplantation activity, university or not, presence of multidisciplinary team. We arbitrarily made a pre-selection of the centers, considering the above questions, to invite to participate of the study. The number of patients per center will be set in relation to the number of patients being followed. Patients will be randomly selected in a regular office visit using routine computerized method previously defined.

Data Collection: Data will be collected in 6-12 months and directly register in the Research Electronic Data Capture (RedCap) system during a regular office visit to transplant service, by a trained professional. The RedCap is a safe internet program, created by the Vanderbilt University, designed exclusively for capture and storage of data that can be powered remotely by trained people. The Federal University of Juiz de Fora is part of the consortium of institutions authorized to use this program. It allows data to be collected, organized and stored in the same action, making the process of data analysis (http://www.project-redcap.org/).

VARIABLES AND MEASUREMENTS

The implementation phase of medication adherence (taking and timing dimensions, drug holidays and dose reduction) to immunosuppressive drugs is measured using three methods: a validated self-report (Basel Assessment of Adherence with Immunosuppressive Medication Scale - BAASIS), blood assay and collateral reports by health care workers.

Non-adherence to immunosuppressive drugs:

1. Self-reported non adherence: It will be measured using the four-item validated self-report The Basel Assessment of Adherence Scale for Immunosuppressive (BAASIS) which was recently validated to Brazilian Portuguese by our group5.
2. Collateral report: In addition, we will use a qualitative method of measuring adherence - the collateral report. We will ask to the nurse and to the medical assistant directly responsible for the follow-up care of the KTx recipients to score patients' adherence in one of three categories: good, fair or poor. "Good" or "fair" answers by one of the professionals classifies the patients as non-adherent.8
3. Blood assay: Patients´ adherence will also measured checking if the trough blood levels of the immunosuppressive drugs are within the therapeutic range.9 Composite adherence score: In order to increase diagnostic accuracy, a composite adherence score will be calculate based on findings of the BAASIS, collateral report and blood assay. Overall NAd will be define as an indication of NAd by one of the three methods.7,8

The current physical activity level (till 150minutes/week of moderate exercise), smoking status (current), alcohol use [(>1 drink/day (women), >2 drinks/day (men)] , and appointment keeping (missed ≥ 1 appointment/last 5) are assessed by using investigator-developed questions based on previous transplant research.

Risk factors of NAd: All the five WHO dimensions will be evaluated: socio-economic (age - years; gender; race - self-defined, white or other; highest level of education; employment; marital status - married or not; family income - per month; patient-related (smoking and alcohol intake - yes,no or social, ability in identifying the immunosuppressants in use); condition/disease-related (time on dialysis - months, dialysis modality - peritoneal or hemodialysis or preemptive transplant, post transplant time - months, previous acute rejection - as recorded in the file, creatinine, actual chronic kidney disease(-CKD) stage, estimated by CKD-EPI study formulae), therapy/treatment-related (donor - deceased, living-related, or living-unrelated donor graft; number of prescribed medications, number of dosing times) and healthcare system/healthcare worker-related factors (city of origin-same or different from transplant´s center, distance to transplant center -in miles, private insurance - yes or no, and subjective evaluation of the health workers (physician and nurse; if satisfied or not). Data will be collected from medical files and directly by a complementary questionnaire.

STATISTICAL PROCEDURES Baseline characteristics will be described as continuous variables as mean ± standard deviation or median with range whenever will appropriate. Categorical variables were represented as frequencies. For checking the normality of the sample, the Kolmogorov-Smirnov and Shapiro-Wilk tests will be conducted. T-Test, Mann-Whitney and Chi-square or Fisher´s Tests will be use to assess association between explanatory variables and adherence status. Multivariate Logistic Regression analysis will be performed to assess the association between the variables on the outcome of adherence. Statistical analysis will be performed using SPSS software v.19.0 for Windows (EUA, Chicago). A p value <0.05 will consider significant.

ELIGIBILITY:
Inclusion Criteria:

* Being at least 18 years old
* More than 1 year posttransplant
* Willing to participate in the study by signing a written informed consent form.

Exclusion Criteria:

- Retransplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney Transplant patient
Sampling Method: Non-Probability Sample
Enrollment: 1105 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
adherence to immunosuppressives | 1 day
  Adherence will be defined by three methods: The BAASIS instrument, blood assay of the immunosuppressives and collateral report. A patients is classified as non-adherent if he/she is considered non-adherent by any of the methods.

SECONDARY OUTCOMES:
Risk factors to non-adherence | 1 day
  Risk factors to non-adherence are socio-economic; patient-related; condition/disease-related; therapy/treatment-related;healthcare system/healthcare worker-related factors

CONTACTS AND LOCATIONS:
Overall Officials: HELADY S PINHEIRO, MD, PhD, Principal Investigator — Fundação Instituto Mineiro de Estudos e Pesquisas em Nefrologia
Locations (1):
- Fundação Instituto Mineiro de Estudos e Pesquisas em Nefrologia, Juiz de Fora, Minas Gerais, Brazil

REFERENCES:
- [Background] Neipp M, Jackobs S, Klempnauer J. Renal transplantation today. Langenbecks Arch Surg. 2009 Jan;394(1):1-16. doi: 10.1007/s00423-008-0335-1. Epub 2008 May 14. PMID 18478256
- [Background] Sabaté E. Adherence to long-term therapies: Evidence for action. Geneva: World Health Organization. 2003.
- [Background] Denhaerynck K, Dobbels F, Cleemput I, Desmyttere A, Schafer-Keller P, Schaub S, De Geest S. Prevalence, consequences, and determinants of nonadherence in adult renal transplant patients: a literature review. Transpl Int. 2005 Oct;18(10):1121-33. doi: 10.1111/j.1432-2277.2005.00176.x. PMID 16162098
- [Background] Michelon TF, Piovesan F, Pozza R, Castilho C, Bittar AE, Keitel E, Santos A, Goldani JC, Garcia CD, Neumann J, Garcia VD. Noncompliance as a cause of renal graft loss. Transplant Proc. 2002 Nov;34(7):2768-70. doi: 10.1016/s0041-1345(02)03403-6. No abstract available. PMID 12431602
- [Background] Marsicano Ede O, Fernandes Nda S, Colugnati F, Grincenkov FR, Fernandes NM, De Geest S, Sanders-Pinheiro H. Transcultural adaptation and initial validation of Brazilian-Portuguese version of the Basel assessment of adherence to immunosuppressive medications scale (BAASIS) in kidney transplants. BMC Nephrol. 2013 May 21;14:108. doi: 10.1186/1471-2369-14-108. PMID 23692889
- [Background] Registro Brasileiro de Transplante 2012 [Online]. Available at: http://www.abto.com.br/profissionais.
- [Background] Osterberg L, Blaschke T. Adherence to medication. N Engl J Med. 2005 Aug 4;353(5):487-97. doi: 10.1056/NEJMra050100. No abstract available. PMID 16079372
- [Background] Schafer-Keller P, Steiger J, Bock A, Denhaerynck K, De Geest S. Diagnostic accuracy of measurement methods to assess non-adherence to immunosuppressive drugs in kidney transplant recipients. Am J Transplant. 2008 Mar;8(3):616-26. doi: 10.1111/j.1600-6143.2007.02127.x. PMID 18294158
- [Background] Denhaerynck K, Burkhalter F, Schafer-Keller P, Steiger J, Bock A, De Geest S. Clinical consequences of non adherence to immunosuppressive medication in kidney transplant patients. Transpl Int. 2009 Apr;22(4):441-6. doi: 10.1111/j.1432-2277.2008.00820.x. Epub 2008 Dec 24. PMID 19144090
- [Derived] Karlburger RL, de Pinho JHS, Basile Colugnati FA, Denhaerynck K, Medina JOP, Veras de Sandes-Freitas T, De Geest S, Sanders-Pinheiro H; ADHERE BRAZIL Study Team. Associated Factors to Nonadherence to Routine Appointments after Kidney Transplantation: The ADHERE Brazil Study. Clin Transplant. 2025 Oct;39(10):e70339. doi: 10.1111/ctr.70339. PMID 41055605
- [Derived] Marsicano-Souza EO, Colugnati FAB, de Castro BBA, Van Keullen MDS, De Geest S, Sanders-Pinheiro H. Management strategies for implementing a multicenter cross-sectional study: lessons from the ADHERE Brazil study. Sao Paulo Med J. 2022 May-Jun;140(3):439-446. doi: 10.1590/1516-3180.2021.0492.R1.15092021. PMID 35507993
- [Derived] Sanders-Pinheiro H, Colugnati FAB, Marsicano EO, De Geest S, Medina JOP; Adhere Brazil Consortium Group. Prevalence and correlates of non-adherence to immunosuppressants and to health behaviours in patients after kidney transplantation in Brazil - the ADHERE BRAZIL multicentre study: a cross-sectional study protocol. BMC Nephrol. 2018 Feb 20;19(1):41. doi: 10.1186/s12882-018-0840-6. PMID 29463231